CLINICAL TRIAL: NCT04726111
Title: COVID-19 and Pregnancy: Placental and Immunological Impacts
Acronym: MaterCov
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020_0170
Record Dates: First submitted 2021-01-21; First posted 2021-01-27 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control patients (Other): Control patients (negative serology and PCR)
  Interventions: Other: Specimens specific for the study
- asymptomatic patients (Other): asymptomatic patients (PCR positive)
  Interventions: Other: Specimens specific for the study
- symptomatic patients (Other): symptomatic patients (PCR positive)
  Interventions: Other: Specimens specific for the study
- Cured patients (Other): cured patients who contracted the disease during pregnancy (positive serology in the 15 days preceding childbirth or history of positive PCR during pregnancy and negative PCR within 72 hours)
  Interventions: Other: Specimens specific for the study

INTERVENTIONS:
Other: Specimens specific for the study — Specimens (blood, umbilical cord, umbilical cord blood, placenta)

SUMMARY:
The aim of this study is to compare placental pathologies in patients with COVID 19 infection at the time of childbirth or a history of COVID 19 during pregnancy versus control patients

DETAILED DESCRIPTION:
The second wave of COVID 19 is currently sweeping through Europe. If the first wave brought reassuring elements on the risk of maternal-fetal transmission, it nevertheless counted an increase in severe maternal forms in the third trimester associated with more premature deliveries and cesarean sections. In addition, due to the very recent nature of this new infection, we have little data on the effect of SARS-COV 2 contracted during pregnancy on the fetus and on maternal-fetal exchanges.

Publications report an increase in growth retardation, maternal coagulopathies, preeclampsia and placental thrombosis. The vascular placental abnormalities observed in the first series must be confirmed and refined. Finally, pregnancy is marked by immunomodulation which can interfere with immune reactions. A better understanding of the immunological mechanisms in the mother and of the immunity transmitted to the fetus is necessary to better understand the maternal-fetal issues of COVID 19.

This prospective study concerns patients presenting for their delivery at Foch Hospital.

4 groups of patients will be identified in the delivery room after childbirth based on their COVID 19 PCR taken within 72 hours, their COVID 19 serology, or a history of positive COVID 19 PCR during pregnancy : 1 control group of 50 patients, 1 group of 50 asymptomatic patients, 1 group of 50 patients with symptoms, and 1 group of 50 cured patients who contracted the disease during pregnancy. The patients will have various samples: blood, umbilical cord blood, umbilical cord, placenta

ELIGIBILITY:
Inclusion Criteria:

* Patient pregnant for more than 20 weeks with amenorrhea
* Having completed a COVID 19 PCR within 72 hours
* Admitted to the birthing room at Foch hospital for her delivery

Exclusion Criteria:

* Minor (age <18 years, on inclusion)
* Diabetes with and without insulin (only for the control group)
* High blood pressure (only for the control group),
* Preeclampsia (only for the control group)
* Infection during pregnancy: HIV, toxoplasmosis, rubella, CMV, syphilis.
* PCR Influenza A or B positive, proven by nasopharyngeal swab in the week preceding childbirth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Placental histological evaluation | Delivery Day 0-Day1
  vascular hypoperfusion on the fetal and maternal side, thrombosis and other abnormalities

SECONDARY OUTCOMES:
Cellular analysis on maternal blood and cord blood: phenotyping from PBMCs and NFS with the characterization of lymphocyte populations by the CytodiffTM technique | Delivery Day 0 - Day 1
Cellular analysis on maternal blood and cord blood: functional activities from PBMCs and NFS with the characterization of lymphocyte populations by the CytodiffTM technique | Delivery Day 0 - Day 1
Number of cytokines in maternal blood and cord blood | Delivery Day 0 - Day 1
Number of immunoglobulins in maternal and fetal blood | Delivery Day 0 - Day 1
Maternal clinical evaluation then neonatal on medical file and telephone questionnaire 1 month after childbirth. Comparison of results between groups. | 1 month postpartum Day 30
  Maternal clinical evaluation (preeclampsia, retroplacental hematoma, severe symptoms of the disease, cesarean section for respiratory distress, hemorrhage during delivery, length of hospitalization, re-hospitalization within 30 days, sequelae) and fetal then neonatal (fetal death in utero , intrauterine growth retardation, premature delivery, birth weight, pH, cord lactates, APGAR score, neonatal hospitalization, intensive care hospitalization, length of hospitalization, notion of COVID 19 infection in the month that following childbirth) based on medical records and telephone questionnaire 1 month after childbirth. Comparison of results between groups.
Foetal clinical evaluation then neonatal on medical file and telephone questionnaire 1 month after childbirth. Comparison of results between groups. | 1 month postpartum Day 30
  Maternal clinical evaluation (preeclampsia, retroplacental hematoma, severe symptoms of the disease, cesarean section for respiratory distress, hemorrhage during delivery, length of hospitalization, re-hospitalization within 30 days, sequelae) and fetal then neonatal (fetal death in utero , intrauterine growth retardation, premature delivery, birth weight, pH, cord lactates, APGAR score, neonatal hospitalization, intensive care hospitalization, length of hospitalization, notion of COVID 19 infection in the month that following childbirth) based on medical records and telephone questionnaire 1 month after childbirth. Comparison of results between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Foch, Suresnes, France